CLINICAL TRIAL: NCT03049384
Title: Tailored Exercise Interventions to Reduce Fatigue in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Guillaume Millet, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-16-1010
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Cancer-related Fatigue

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Exercise (Active Comparator): A classical exercise intervention based on current guidelines for cancer survivors.
  Interventions: Other: Traditional Exercise
- Tailored Exercise (Experimental): A tailored and individualized exercise intervention based on the results of pre-intervention testing.
  Interventions: Other: Tailored Exercise

INTERVENTIONS:
Other: Traditional Exercise — The traditional exercise group will undertake a supervised exercise intervention involving aerobic exercise and light resistance training, in line with published guidelines for exercise in cancer survivors.
  Arms: Traditional Exercise
Other: Tailored Exercise — The tailored training group will be prescribed an individualized exercise intervention designed specifically to counteract deficits (e.g. neuromuscular) of difficulties (e.g. sleep disturbance) identified during pre-intervention testing.
  Arms: Tailored Exercise

SUMMARY:
Cancer-related fatigue (CRF) is a common and distressing symptom of cancer and/or cancer treatment that can persist for months or years in cancer survivors. Exercise is beneficial for the management of CRF, and general exercise guidelines for cancer survivors are available. However, exercise interventions have not been tailored to alleviate CRF in fatigued cancer survivors, and thus the potential to alleviate CRF may not have been realized. The primary aim of this research is to investigate the effect of a traditional vs. tailored 12-week exercise intervention on self-reported CRF severity.

DETAILED DESCRIPTION:
Background and Rationale

Approximately one-third of cancer survivors experience severe and persistent fatigue for a number of years post-treatment, but this distressing symptom is often under-treated by healthcare professionals due to a lack of mechanism-targeted interventions. The assessment of cancer-related fatigue (CRF) is reliant on subjective fatigue measurements such as self-report questionnaires. Less attention has been given to objective physiological measurements. However, there are well-established techniques which allow the assessment of neuromuscular fatigue and its peripheral and central origins which could be utilized in the study of CRF. Very few studies have considered these objective measures alongside self-report scales in the study of CRF and only two have used such techniques in cancer survivors. To date, no studies have investigated neuromuscular fatigue in whole body, dynamic activity as relevant to daily tasks (and involving the lower limb due to its functional relevance to locomotion). Novel testing developed in our laboratory could be used as part of a wider screening to develop individualized interventions to alleviate CRF. It is well accepted in the field that CRF is multidimensional and in addition to a potential neuromuscular component, the role of sleep disturbance may also be implicated. Interventions targeted at improving sleep quality are therefore warranted, and there is sound evidence for the efficacy of exercise interventions in particular for improving CRF in cancer survivors. As a non-pharmacological intervention, physical activity has the strongest evidence base for treating CRF. However, the mechanisms explaining the reduction of CRF with exercise are not understood. Due to the complex and multi-factorial nature of CRF, it would be of benefit to tailor exercise interventions to the specific deficits (in regards to neuromuscular mechanisms) or difficulties (for example sleep disturbance) experienced by the individual. Ultimately, mechanism-targeted exercise interventions could be translated to clinical rehabilitation programs and lead to an improved quality of for cancer survivors.

Research Question & Objectives

The primary aim of this research is to investigate the effect of a traditional vs. tailored 12-week exercise intervention on self-reported CRF severity.

Methods

Fatigued cancer survivors who have completed primary treatment ≥ 3 months and ≤ 5 years from enrollment will be randomly allocated to one of two treatment arms: traditional (active control) and tailored exercise. Participants in the traditional exercise group will engage in aerobic and resistance exercise that is consistent with published recommendations. The tailored exercise group will be prescribed an intervention designed to address individual deficits (identified at baseline) that may be related to CRF. Participants will be assessed before and after the intervention for patient-reported outcomes, neuromuscular function and fatigue in response to whole-body exercise, sleep quantity and quality, physical activity levels, cardiorespiratory fitness and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years;
* Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score ≤ 34;
* Completion of treatment in ≥ 3 months and ≤ 5 years preceding enrollment;
* Approval received from personal physician and/or a Canadian Society for Exercise Physiology-Clinical Exercise Physiologist (CSEP-CEP);
* Command of the English language.

Exclusion Criteria:

* Contraindication to experimental procedures including transcranial magnetic stimulation (TMS);
* Diagnosed as having obstructive sleep apnea or anemia;
* Currently participating in a structured exercise intervention;
* Participant is pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Scale | Baseline to after the 12-week intervention, at 6 month and 12 month follow up.
  Self-report questionnaire for the assessment of cancer-related fatigue.

SECONDARY OUTCOMES:
Assessment of change in The Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline and after the 12-week intervention.
  General quality of life instrument intended for use with a variety of chronic illness conditions.
Assessment of change in Edmonton Symptom Assessment System-revised tiredness scale | Baseline and after the 12-week intervention, and during follow up (6 and 12 months).
  Self-report questionnaire for the assessment of of nine common symptoms experienced by cancer patients.
Maximal Isometric Force in the Knee Extensors | Baseline and after the 12-week intervention.
  A reduction in maximal isometric force in the knee extensors measured before, during and after an intermittent cycling test.
Cortical Voluntary Activation | Baseline and after the 12-week intervention.
  A reduction voluntary activation (using transcranial magnetic stimulation) measured measured before, during and after an intermittent cycling test.
Voluntary Activation | Baseline and after the 12-week intervention.
  A reduction voluntary activation (using femoral nerve stimulation) measured before, during and after an intermittent cycling test.
Potentiated Doublet Twitch Force | Baseline and after the 12-week intervention.
  A reduction in potentiated quadriceps twitch force (from a high frequency doublet at 100 Hz) measured before, before, during and after an intermittent cycling test.
Muscle Compound Action Potential (M-Wave) Peak-to Peak Amplitude | Baseline and after the 12-week intervention.
  Evoked from supra-maximal stimulation of the femoral nerve and measured before, during and after an intermittent cycling test.
Muscle Compound Action Potential (M-Wave) Peak-to Peak Duration | Baseline and after the 12-week intervention.
  Evoked from supra-maximal stimulation of the femoral nerve and measured before, during and after an intermittent cycling test.
Muscle Compound Action Potential (M-Wave) Area | Baseline and after the 12-week intervention.
  Evoked from supra-maximal stimulation of the femoral nerve and measured before, during and after an intermittent cycling test.
Motor Evoked Potential (MEP) Peak-to Peak Amplitude | Baseline and after the 12-week intervention.
  Normalized to the maximal M-wave and measured before, during and after an intermittent cycling test.
Motor Evoked Potential (MEP) Peak-to Peak Duration | Baseline and after the 12-week intervention.
  Normalized to the maximal M-wave and measured before, during and after an intermittent cycling test.
Motor Evoked Potential (MEP) Area | Baseline and after the 12-week intervention.
  Normalized to the maximal M-wave and measured before, during and after an intermittent cycling test.
Cortical Silent Period | Baseline and after the 12-week intervention.
  Evoked from TMS and measured (from stimulation artifact to the continuous resumption of EMG) before, during and after an intermittent cycling test.
Voluntary Electromyography (EMG) | Baseline and after the 12-week intervention.
  Root mean square of the EMG signal during an MVC, measured before, during and after an intermittent cycling test.
Amplitude of the Sleep-Wake Cycle | Baseline and after the 12-week intervention.
  The mean difference between lowest and highest activity period, recorded with actigraphy.
Peak Time of the sleep-wake Cycle | Baseline and after the 12-week intervention.
  Time of day of the highest estimated level of wake, recorded by actigraphy.
Mesor of the Sleep-Wake Cycle | Baseline and after the 12-week intervention.
  Mean level of activity over 24 hours, recorded with actigraphy.
inter-daily stability | Baseline and after the 12-week intervention.
  the degree of regularity of the rest-activity patterns on individual days in the 24 h environment, recorded with actigraphy.
intra-daily variability | Baseline and after the 12-week intervention.
  the fragmentation of periods of rest and activity, recorded with actigraphy.
L5 | Baseline and after the 12-week intervention.
  The mean activity counts in the least active 5 h period in the average 24 h pattern) recorded with actigraphy.
L5 mid | Baseline and after the 12-week intervention.
  The central time of the L5 period, usually referring to the through of the activity period), recorded with actigraphy.
Wake actigraphy | Baseline and after the 12-week intervention.
  Amount of activity during wake, recorded with actigraphy
Sleep Activity | Baseline and after the 12-week intervention.
  Amount of activity during sleep periods, recorded with actigraphy
Activity Index | Baseline and after the 12-week intervention.
  Percentage of activity per epoch for wake and sleep, recorded with actigraphy.
Time in bed | Baseline and after the 12-week intervention.
  Time spent between the moment subject turn off the light to sleep and the moment he gets up, recorded with actigraphy.
Actual Sleep Time | Baseline and after the 12-week intervention.
  Time spent asleep during the night, recorded with actigraphy.
Actual Wake Time | Baseline and after the 12-week intervention.
  Time spent awaken during the night, recorded with actigraphy.
Sleep Onset Latency | Baseline and after the 12-week intervention.
  Time to fall asleep, recorded with actigraphy.
Sleep Efficiency | Baseline and after the 12-week intervention.
  Ratio between the time spent asleep and the total duration of sleep period, recorded with actigraphy.
Fragmentation index | Baseline and after the 12-week intervention.
  Indication of the sleep quality based on movement during night, recorded with actigraphy.
Blood Biomarkers | Baseline and after the 12-week intervention.
  Blood count, catecholamines, serotonin, cortisol, inflammatory markers and markers of oxidative stress.
Assessment of change in the Centre for Epidemiological Studies Depression Scale (CES-D) questionnaire. | Baseline and after the 12-week intervention.
  Self-report questionnaire for the assessment of health-related quality of life, specific to cancer type.
Assessment of change in The Social Prevision Scale (SPS) | Baseline and after the 12-week intervention.
  Self-report questionnaire for the assessment of social support.
Assessment of change in The Functional Assessment of Cancer Therapy (FACT) Cancer Specific | Baseline and after the 12-week intervention.
  Self-report questionnaire for the assessment
Assessment of change in The Modified-Godin Leisure Time Exercise Questionnaire (GLTEQ) | Baseline, after the 12-week intervention, and during follow up (6 and 12 months).
  Self-report questionnaire for the assessment of leisure time physical activity.
Assessment of change in The Insomnia Severity Index (ISI) | Baseline and after the 12-week intervention.
  Self-report questionnaire for the assessment of insomnia severity.
Assessment of change in The Brief Pain Inventory Short Form (BPI-sf) | Baseline and after the 12-week intervention.
  Self-report questionnaire for the assessment of pain.
Assessment of change in Maximal Oxygen Uptake | Baseline and after the 12-week intervention.
  The highest 30 second average oxygen uptake measured during an an incremental cycling test.
Assessment of change in Muscle Cross-Sectional Area | Baseline and after the 12-week intervention.
  Ultrasound measurement of the vastus lateralis and rectus femoris.
Heart Rate Variability | Baseline and after the 12-week intervention.
  Variation in the time interval between heartbeats.
Assessment of change in Fat Mass | Baseline and after the 12-week intervention.
  Measured using dual energy X-ray absorptiometry (DXA).
Assessment of change in Fat Free Mass | Baseline and after the 12-week intervention.
  Measured using dual energy X-ray absorptiometry (DXA).
Assessment of change in Bone Mineral Density | Baseline and after the 12-week intervention.
  Measured using dual energy X-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Millet, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Twomey R, Martin T, Temesi J, Culos-Reed SN, Millet GY. Tailored exercise interventions to reduce fatigue in cancer survivors: study protocol of a randomized controlled trial. BMC Cancer. 2018 Jul 24;18(1):757. doi: 10.1186/s12885-018-4668-z. PMID 30041626